CLINICAL TRIAL: NCT04370392
Title: Intraperitoneal Versus Intravenous Dexmedetomidine for Post-operative Analgesia Following Laparoscopic Sleeve Gastrectomy Surgery, A Prospective Randomized Control Trial.
Brief Title: Intraperitoneal Versus Intravenous Dexmedetomidine for Post-operative Analgesia Following Laparoscopic Sleeve Gastrectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IV and IP detomidinemidine
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Postoperative Pain After Laparoscopic Sleeve Gastrectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): intraperitoneal local anesthetic instillation (40 ml bupivacaine 0.25%) through the trocar with intravenous infusion of 50 ml normal saline over 10 minutes.
  Interventions: Procedure: intraperitoneal local anaesthetic instillation
- IV dexmedetomidine group (Experimental): intraperitoneal local anesthetic instillation (40 ml bupivacaine 0.25%) through the trocar with intravenous infusion of 50 ml normal saline containing dexmedetomidine 1 ug/kg over 10 minutes.
  Interventions: Procedure: intraperitoneal local anaesthetic instillation
- IP dexmedetomidine group (Experimental): intraperitoneal anesthetic instillation (40 ml total volume containing bupivacaine 0.25% with dexmedetomidine 1 ug/kg) through the trocar with intravenous infusion of 50 ml normal saline over 10 minutes.
  Interventions: Procedure: intraperitoneal local anaesthetic instillation

INTERVENTIONS:
Procedure: intraperitoneal local anaesthetic instillation — intraperitoneal anesthetic instillation (40 ml total volume containing bupivacaine 0.25) through the trocar at the subdiaphragmatic space in Trendelenburg's position for 5 min with intravenous infusion of 50 ml normal saline over 10 minutes.

SUMMARY:
One of most common bariatric surgery is laparoscopic sleeve gastrectomy. Pain after laparoscopic surgery may be due to stretching of the intra-abdominal cavity, peritoneal inflammation, and diaphragmatic irritation caused by residual carbon-dioxide in the peritoneal cavity.Multimodal efforts like parenteral opioids, non-steroidal anti-inflammatory drugs or local wound infiltration have been done to reduce overall pain and benefit post-operative conditions of patients undergoing laparoscopic surgeries. Despite their efficacy, with all parenteral medications, there are associated adverse effects.

Intraperitoneal local anesthetic is a safe and effective analgesic approach which used to control pain after laparoscopic surgery. Many authors have evaluated the role of IP local anesthetic administration in laparoscopic colorectal cancer surgery, laparoscopic cholecystectomy, laparoscopic appendectomy and laparoscopic hysterectomy

DETAILED DESCRIPTION:
Laparoscopic procedures have many advantages over open procedures such as lesser haemorrhage, better cosmetic results, lesser post-operative pain, and shorter recovery time, leading to shorter hospital stay and less expenditure.One of most common bariatric surgery is laparoscopic sleeve gastrectomy. Pain after laparoscopic surgery may be due to stretching of the intra-abdominal cavity, peritoneal inflammation, and diaphragmatic irritation caused by residual carbon-dioxide in the peritoneal cavity.

Multimodal efforts like parenteral opioids, non-steroidal anti-inflammatory drugs or local wound infiltration have been done to reduce overall pain and benefit post-operative conditions of patients undergoing laparoscopic surgeries. Despite their efficacy, with all parenteral medications, there are associated adverse effects.

Intraperitoneal local anesthetic is a safe and effective analgesic approach which used to control pain after laparoscopic surgery. Many authors have evaluated the role of IP local anesthetic administration in laparoscopic colorectal cancer surgery, laparoscopic cholecystectomy, laparoscopic appendectomy and laparoscopic hysterectomy.

Dexmedetomidine (alpha-2 adrenergic agonists) has become one of the frequently used drugs in anesthesia as it has been reported to provide analgesia, anxiolysis, and an anesthetic-sparing action with minimal respiratory depression plus its sedative effect that mimics natural sleep. Dexmedetomidine can used safely both intravenous and plus bupivacaine in different nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic sleeve gastrectomy who meet the known criteria for bariatric procedures (BMI ≥ 40 or 35 with comorbidities related to obesity or obesity for more than 5 years with all efforts to reduce weight failing).

Exclusion Criteria:

* 1. Cardiac patients, 2. patients with known allergy to bupivacaine, 3. prolonged administration of NSAIDS or other analgesics due to chronic pain of any reason, 4. severe renal and hepatic diseases, 5. on antihypertensive medication with any α2 adrenergic agonists, e.g., clonidine or beta blockers 6. heart block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Time of first analgesic request | postoperative first day
  Time of first analgesic request when visual analogue score more than 3

SECONDARY OUTCOMES:
postoperative pain assessment | postoperative first day
  Assessment of postoperative pain with Visual analogue scale
Total amount of rescue analgesia | postoperative first day
  Total amount of rescue tramadol analgesia
Number of patients who needed postoperative rescue analgesia | postopertive first day
  Number of patients who needed postoperative rescue tramadol analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Tarek Abdel Hay, Tanta, El Gharbyia, Egypt